CLINICAL TRIAL: NCT01924026
Title: Neuropsychological and Quality of Life Outcomes in Untreated Adults With Mild Hyperphenylalaninemia (MHP)/Phenylketonuria (PKU) With Phenylalanine Levels Between 360 and 600 µmol/L Caused by Phenylalanine Hydroxylase (PAH) Deficiency.
Brief Title: Neurocognitive Outcomes in Mild Hyperphenylalaninemia (MHP)MHP Study
Status: Completed | Type: Observational
Sponsor: The Hospital for Sick Children (Other)
Collaborators: BioMarin Pharmaceutical (Industry)
Responsible Party: Principal Investigator, Annette Feigenbaum, Staff Physician, Metabolic Program, Clinical and Metabolic Genetics, The Hospital for Sick Children
Other Study IDs: 1000039726
Record Dates: First submitted 2013-05-15; First posted 2013-08-16 (Estimated); Last update posted 2016-02-17 (Estimated); Status verified 2016-02

CONDITIONS: Phenylketonuria; Mild Hyperphenylalaninemia
Keywords: Phenylketonuria; Mild Hyperphenylalaninemia; PKU; MHP
MeSH Terms: conditions — Phenylketonurias

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Affected MHP: With Phe between 360 and 600 micromoles/L
- Unaffected Siblings: With normal Phe levels

SUMMARY:
Phenylketonuria (PKU) is a genetic disorder known to cause severe reduction in intelligence and deficits in cognitive function; it is associated with an elevated level of Phenylalanine (Phe) in blood.

Newborn screening and early treatment with restricted protein diet supplemented by a formula of amino-acids will preserve intelligence. In those with the severe form treated from birth, some deficits that affect higher functions of the brain are seen.

Given this, there is disagreement about how milder forms of this disease should be managed and what level of Phe is safe to be left untreated.

We seek to assess whether higher Phe levels, between 360 and 600µmol/L, are safe with respect to preservation of intelligence and higher cognitive functions.

DETAILED DESCRIPTION:
The following personal/medical information will be collected and reviewed:

* Evaluation of current and past medical history, including psychological treatment such as medication and counseling/therapy.
* Mutational analysis for each MHP subject
* Detailed history of educational, employment, relationship, and socioeconomic status/achievements as a measure of successful transition to adulthood
* Diet history, including past treatment with medical food or Sapropterin (Kuvan) for pre-conceptual and pregnancy Phe management
* All available untreated Phe levels, including newborn screening results (where possible) will be collated to calculate lifetime mean Phe level. Age at collections will be recorded separately for each MHP subjects to ensure inclusion of Phe levels beyond infancy

The following clinical investigations will be administered:

* Measurement of Phe and Tyrosine after an overnight fast, via blood spot using tandem mass spectrometry analysis. Blood spot collection will be done at the same time of day for all subjects.
* Physical exam, height and weight measurements
* Food Frequency Questionnaire assessment to estimate typical daily intake of natural protein.
* Self-Report Questionnaires:

  * Behavior Rating Inventory of Executive Function (BRIEF)-A
  * Beck Anxiety Inventory
  * Beck Depression Inventory
  * Quality of Life questionnaire
* Neuropsychological Tests assessed by a trained psychologist

An informant BRIEF-A report will be completed for each subject. To ensure consistency in rating, the same informant will be used where possible for the MHP subject and their sibling control (i.e. parents). These questionnaires will be mailed to the informants and returned to the study site via FedEx.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female, ≥ 18 years
* Confirmed to have MHP with at least two Phe levels during lifetime of above 360µmol/L and below 600µmol/L, including newborn screening levels (available since 1968 by either bacterial inhibition, enzymatic or tandem mass spectrometry methodology) and via mutation analysis. Those with occasional levels above 600µmol/L will not be excluded provided the majority of available levels fall within the 360-600µmol/L range.
* On an unrestricted diet and not taking medical food. Women who were on dietary or Kuvan® treatment for past pre-conception or pregnancy management will not be excluded
* Willing and able to give consent and comply with study procedures.

Exclusion Criteria:

* Subjects on dietary or Kuvan® treatment within the last 12 weeks will be excluded.
* Co-morbidities that may interfere with study participation and/or put the subject at a higher risk of adverse effects.

Subjects who do not have an unaffected sibling may still participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Those with mild form of PKU known as mild hyperphenylalaninemia (MHP) and their unaffected siblings who fulfill the inclusion and exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2013-09; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Executive function | Day 1
  As measured by subtests in Weschler-IV test, and supplemented with assessments from BRIEF-A and CANTAB(computerised cognitive tests by Cambridge Cognition).

SECONDARY OUTCOMES:
Quality of Life | Day 1
Presence of anxiety and depression | Day 1
  As measured by Beck Anxiety and Depression Inventories

OTHER OUTCOMES:
IQ | Day 1
  As measured by Wechsler-IV

CONTACTS AND LOCATIONS:
Overall Officials: Annette Feigenbaum, MD, Principal Investigator — The Hospital for Sick Children; Komudi Siriwardena, MD, Principal Investigator — Stollery Children's Hospital
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
in progress- to be decided.